CLINICAL TRIAL: NCT03776708
Title: What is the Regional and Remote Effect of Spinal Manipulation on Pressure Pain Threshold in Asymptomatic Subjects Over Time: A Randomized Placebo-controlled Study
Brief Title: Effect of Spinal Manipulation on Experimental Pain in Asymptomatic Subjects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Franco Europeen de Chiropratique (Other)
Responsible Party: Principal Investigator, Margaux Honoré, Principal investigator, Institut Franco Europeen de Chiropratique
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: InstitutFEC
Record Dates: First submitted 2018-10-11; First posted 2018-12-17 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Spinal Manipulation
Keywords: pressure pain threshold; asymptomatic subjects; duration
MeSH Terms: interventions — Manipulation, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal manipulation (Experimental): The spinal manipulation is located between the fifth and eighth thoracic vertebrae, on a level and a side pain-free to a light palpation. The maneuver is of high velocity and low amplitude, oriented posterior to anterior, on the transverse process area of the chosen thoracic vertebrae.
  Interventions: Other: Spinal manipulation
- Sham procedure (Sham Comparator): The sham procedure is a manual contact on both inferior angles of the scapulae by the chiropractor. After a short tensioning, a slight movement with low velocity and low amplitude is done, respecting scapula-thoracic sliding plans laterally, without repercussion on the spine. It is considered by us to be a "credible" sham procedure, as it resembles an actual act of thoracic manipulation, and it has been validated, with questionnaires.
  Interventions: Other: Sham procedure

INTERVENTIONS:
Other: Spinal manipulation — Spinal manipulation is defined as a quick, passive and forced manoeuvre applied to spinal joints, and sometimes followed by a characteristic cracking sound. It can be compared to a mobilisation, which is a passive manual therapy as well, but is applied slower and repetitively on the joints. Spinal manipulation has been shown to have a significant clinical impact in the treatment of musculoskeletal pain
  Other Names: Spinal manipulative therapy; Adjustment
  Arms: Spinal manipulation
Other: Sham procedure — The sham procedure is a manual contact on both inferior angles of the scapulae by the chiropractor. After a short tensioning, a slight movement with low velocity and low amplitude is done, respecting scapula-thoracic sliding plans laterally, without repercussion on the spine. It is considered by us to be a "credible" sham procedure, as it resembles an actual act of thoracic manipulation, and it has been validated, with questionnaires
  Other Names: Placebo procedure
  Arms: Sham procedure

SUMMARY:
Spinal manipulation is often used for its effect on pain, but more information is needed concerning its mechanisms of action.

DETAILED DESCRIPTION:
The effect of spinal manipulation on the pressure pain threshold in asymptomatic subjects should be challenged by a validated sham procedure, regionally and remotely over time. Further information is needed concerning its duration and its size.

Research questions:

1. What is the regional effect of spinal manipulation on the pressure pain threshold in asymptomatic subjects, when compared to a valid sham procedure?
2. What is the remote effect of spinal manipulation on the pressure pain threshold in asymptomatic subjects, when compared to a valid sham procedure?
3. What is the duration of the effect of spinal manipulation on the pressure pain threshold in asymptomatic subjects?
4. What is the size of the effect of spinal manipulation on the pressure pain threshold in asymptomatic subjects over time?

ELIGIBILITY:
Inclusion Criteria:

* The subjects must be young (18-30 years old)
* asymptomatic (no pain in the tested area, but the study accepts pain elsewhere, as long as it is less than 1/10 on the BOX-scale).
* Chiropractic students.

Exclusion Criteria:

* The subjects must not be reporting any spinal pain lasting more than a month
* and/or having taken painkillers 24h prior to the study.
* Contra-indications to the spinal manipulation (instability, fracture, malformation, bone or ligament fragility, and inflammations).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Change of the Pressure Pain threshold | The change of the Pressure Pain Threshold is assessed from baseline to immediately after spinal manipulation, and then every fifteen minutes for about an hour.
  Pressure Pain Threshold is defined as the minimal pressure that provokes a pain or a discomfort. It is considered as a valid and objective method, with a good reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Leboeuf-Yde, DC, MPH, PhD, Professor, Study Director — Institut Franco Européen de Chiropraxie
Locations (1):
- Institut Franco Européen de chiropraxie (iFEC), Ivry-sur-Seine, Val De Marne, France